CLINICAL TRIAL: NCT04666363
Title: Evaluation of the Effectiveness of Long-term Inhaled Lavender Applied to Hemodialysis Patients on Invasive Pain Experienced During Cannulation, Patient Comfort, and Anxiety
Brief Title: Inhaled Lavender Applied at Hemodialysis Patients and Effect on Pain, Comfort, and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Demiroglu Bilim University (Other)
Responsible Party: Principal Investigator, Nurten Ozen, Associate Professor, Istanbul Demiroglu Bilim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20978
Record Dates: First submitted 2020-12-08; First posted 2020-12-14 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Hemodialysis
MeSH Terms: interventions — lavender oil

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lavender oil (Experimental): On the first day (before intervention), the intensity of needle insertion-related pain was measured. The experimental group inhaled lavender essence (12 consecutive hemodialysis seasons).
  Interventions: Other: Lavender oil
- Control group (No Intervention): The patients will not smell lavender oil.

INTERVENTIONS:
Other: Lavender oil — the essence was diluted 1:10 with sweet almond oil. A cotton ball soaked in 3 drops of diluted lavender essence was kept at a 10 cm distance from the patients' nose and they were asked to breathe slowly for 5 min.
  Arms: Lavender oil

SUMMARY:
The procedure of puncturing during needle insertion and moving needles within the tissues, the insertion angle, diameter of needles, and insertion techniques all lead the patient to experience pain. However, patients tolerate needle insertion more easily when the pain is managed well. Therefore, pharmacological and non-pharmacological methods are needed in pain control in order to improve comfort when undergoing hemodialysis (HD), and to facilitate patient's compliance to treatment over a longer period. Being one of the non-pharmacological practices, aromatherapy is a part of phototherapy, which means "therapy with plants" and also aims to manage symptoms such as pain as well as the treatment itself.

DETAILED DESCRIPTION:
Experience of the arteriovenous fistula puncture-related pain can have unpleasant effects on the patients, it causes that hemodialysis patients experience more disability, depression, irritability, and insomnia than other patients in adapting to stress. Experiencing continued pain can also affect the level of hemodialysis acceptance in patients and ultimately decrease quality of life. Therefore, pain control is an important priority in these patients. In this regard, in various studies, different pharmacological and non-pharmacological approaches have been used to alleviate the pain.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* On maintenance hemodialysis three times per week for four hours per session
* Receiving hemodialysis therapy for a least six moths at the time of the study
* Having the ability to smell
* Able to communicate in Turkish
* Willing to participate to the study

Exclusion Criteria:

* 18 years of age younger
* Absence of psychiatric disorders that cause cognitive dysfunction, such as Alzheimer's disease or chronic psychosis
* Pregnant women, patients with a history of allergies, respiratory diseases, neuropathy and peripheral vascular diseases
* Administered with painkillers in the past 3 hours
* Having infection at the fistula area
* Requiring more than one attempt for fistula puncturing
* Unwilling to to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline invasive pain at one month | Baseline and one month (At the end of the between 1st and12th dialysis session (3 hemodialysis sessions are done every week))
  It will be assessed at the end of the dialysis session with Visual Analogue Scale. Pain intensity measured on a Visual Analog Scale with scores ranging from 0 - 10. The high point describes bad outcome
Change from baseline comfort at one month | Baseline and one month (At the end of the between 1st and12th dialysis session (3 hemodialysis sessions are done every week))
  It will be assessed first dialysis session and at the end of the 12th dialysis session by the nurse. The lowest point is one, the highest point is five. The high point describes good comfort
Change from baseline anxiety at one month | Baseline and one month (At the end of the between 1st and12th dialysis session (3 hemodialysis sessions are done every week))
  It will be assessed with Hospital Anxiety and Depression Scale. This scale, which has a two-factor structure is comprised of 14 items. Seven of these items assess the anxiety status and the remaining seven assess depression.
  Each item is scored on a four-point scale. Total score ranges between 0 and 21 for anxiety and depression. Scores between 0 and 7 indicate normal emotional status.

CONTACTS AND LOCATIONS:
Locations (1):
- Demiroglu Bilim University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jafari-Koulaee A, Moosazadeh M, Bagheri Nesami M, Goudarzian AH. Effect of cryotherapy on arteriovenous fistula puncture-related pain in hemodialysis patients: A systematic review and meta-analysis. Complement Ther Med. 2020 Mar;49:102326. doi: 10.1016/j.ctim.2020.102326. Epub 2020 Jan 22. PMID 32147063
- [Background] Bouya S, Ahmadidarehsima S, Badakhsh M, Balouchi A, Koochakzai M. Effect of aromatherapy interventions on hemodialysis complications: A systematic review. Complement Ther Clin Pract. 2018 Aug;32:130-138. doi: 10.1016/j.ctcp.2018.06.008. Epub 2018 Jun 13. PMID 30057040
- [Background] Lakhan SE, Sheafer H, Tepper D. The Effectiveness of Aromatherapy in Reducing Pain: A Systematic Review and Meta-Analysis. Pain Res Treat. 2016;2016:8158693. doi: 10.1155/2016/8158693. Epub 2016 Dec 14. PMID 28070420